CLINICAL TRIAL: NCT03011177
Title: A Randomized, Open Label, Parallel-group, Non-inferiority, Active-controlled, Phase Ⅳ Study to Evaluate the Efficacy and Safety of Teneligliptin Versus Linagliptin in Type 2 Diabetes Mellitus Patients
Brief Title: Teneligliptin Versus Linagliptin in Diabetes Mellitus Type Two Patients
Acronym: TELIUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP_C402
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Type2 Diabetes Mellitus
MeSH Terms: interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Linagliptin

ARMS (2):
- teneligliptin (Experimental): teneligliptin 20mg qd
  Interventions: Drug: Teneligliptin
- linagliptin (Active Comparator): linagliptin 5mg qd
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: Teneligliptin — teneligliptin 20mg qd
  Arms: teneligliptin
Drug: Linagliptin — linagliptin 5mg qd
  Arms: linagliptin

SUMMARY:
To assess the efficacy and safety of Teneligliptin and Linagliptin in the type 2 Diabetes Mellitus patients.

DETAILED DESCRIPTION:
A randomized, open label, parallel-group, non-inferiority, active-controlled, phase IV study

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 19 years or older on screening
* Patients with type 2 diabetes mellitus
* Patients with 7.0% ≤ HbA1c ≤ 11.0% at the screening visit
* Patients with Fasting Plasma Glucose <15mmol/L(270mg/dL) on screening

Exclusion Criteria:

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12week

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea